CLINICAL TRIAL: NCT07290530
Title: A 24-Month, Randomized, Double-Masked, Placebo-Controlled Trial of NPI-001 for the Preservation of Photoreceptors in Retinitis Pigmentosa Associated With Usher Syndrome
Brief Title: 24-Month Trial of NPI-001 for the Preservation of Photoreceptors in Retinitis Pigmentosa Associated With Usher Syndrome
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nacuity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-24-01
Record Dates: First submitted 2025-12-16; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Retinitis Pigmentosa (RP); Usher Syndrome
Keywords: N-acetylcysteine amide
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes | interventions — N-Acetylcysteinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NPI-001 (Experimental): NPI-001 tablet, BID
  Interventions: Drug: N-acetylcysteine amide
- Placebo (Placebo Comparator): Placebo tablet, BID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine amide — N-acetylcysteine amide (NPI-001) tablets (250 mg), taken BID
  Arms: NPI-001
Other: Placebo — Placebo tablets, BID
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if NPI-001 works to prevent progression of retinitis pigmentosa in adults diagnosed with Usher syndrome. It will also provide information about the safety of NPI-001. The main questions it aims to answer are:

Does NPI-001 slow down the loss of photoreceptors? What medical problems do participants have when taking NPI-001? Researchers will compare NPI-001 to a placebo (a look-alike substance that contains no drug) to see if NPI-001 works to preserve vision.

Participants will:

Take NPI-001 or a placebo twice a day, every day for 24 months Visit the clinic 9 times for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form (ICF) and to adhere to the study protocol.
2. Diagnosed with Usher syndrome.
3. EZ zone width ≥ 500 microns, which includes the fovea in each eye at Visit 1 (Screening).
4. All edges of the EZ area in both eyes can be visualized at Visit 1 (Screening).
5. Have at least 20 detectable points on the MAIA grid in at least one eye at the Screening and Baseline visits (same eye for both visits).

5. On stable dose of medications associated with other conditions for at least one month.

6. Both female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a bilateral oophorectomy, hysterectomy or bilateral salpingectomy; must abstain from intercourse; or must agree to practice 2 acceptable methods of contraception throughout the course of the study and 4 weeks after the last visit. Acceptable methods of contraception include hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods (diaphragm, condom) with spermicide, tubal ligation, and vasectomy.

Exclusion Criteria:

1. Concurrent retinal pathologies that result in vision loss or inability to fixate, including but not limited to, choroideremia, retinal vein occlusion, and neovascular age-related macular degeneration.
2. Intraocular surgery within the last two months or capsulotomy within the last month.
3. Current or history of uveitis, Coat's disease, diabetic retinopathy, glaucoma, herpes simplex of the eye, or currently has a cataract that prevents visualization of the posterior pole.
4. Likely to require cataract surgery within the next 12 months.
5. Unstable fixation during microperimetry in either eye at either Screening or Baseline visits.
6. Use of any other investigational new drug, or participation in another clinical trial within 12 weeks before the start of study treatment.
7. Use of N-acetylcysteine containing products in the previous 30 days prior to the baseline visit or unwilling to refrain from such supplements for the duration of the study.
8. Chronic liver or kidney disease, cystic fibrosis, severe asthma, or chronic obstructive pulmonary disease (COPD), history of thrombocytopenia not due to a reversible cause, or other blood dyscrasia.
9. Suspected liver dysfunction determined by having alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin values > 1.5 X the upper limit of normal (ULN) at screening.
10. Platelet or hemoglobin values < 100 at screening.
11. History of known sensitivity to N-acetylcysteine or similar thiol compounds or any ingredients of NPI-001.
12. History of hypersensitivity to any medication or food resulting in systemic symptoms.
13. History of cancer (other than non-melanoma skin cancer) diagnosed or requiring treatment within the past 2 years.
14. Pregnant women or women planning to become pregnant in the next 25 months or men with partners planning to become pregnant in the next 25 months.
15. Lactating women who are breast-feeding.
16. Potential participant lives in the same household as a current participant in this study.
17. Subjects who are willing or unable to refrain from donation of blood from 30 days prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening until 56 days following the last study drug dose administered.
18. Inability to provide blood samples, including difficulty with venous access.
19. Any reason, in the opinion of the Principal Investigator, the participant should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
EZ Area Rate of Change | 24 months

IPD SHARING:
Plan to Share IPD: Undecided